CLINICAL TRIAL: NCT05807880
Title: The First-line Therapy With the Combination of Anlotinib, Penpulimab and Capecitabine in Recurrent/Metastatic Nasopharyngeal Carcinoma: a Single-arm, Open-label, Phase II Trial
Brief Title: Anlotinib, Penpulimab and Capecitabine in Recurrent/Metastatic Nasopharyngeal Carcinoma
Acronym: ALTER-HN005
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-HN005
Record Dates: First submitted 2023-03-28; First posted 2023-04-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — penpulimab; Capecitabine

STUDY DESIGN:
Intervention Model Description: The combination of anlotinib, penpulimab and capecitabine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): First, patients will receive the combination treatment of anlotinib, penpulimab and capecitabine every three weeks for 4-6 cycles. For each cycle, patients receive anlotinib 10mg, po, qd from day 1 to day 14, penpulimab 200mg, iv in day 1, and capecitabine 650mg/m2, po, bid from day 1 to day 21. Then a maintenance treatment will be run with "penpulimab and capecitabine"(the dose and the medication method remain the same) for every 3 weeks until PD or intolerance to drug toxicity.
  Note: After using the penpulimab for 2 years, it is dependent on the researcher's judgement of the benefit evaluation whether to continue using it.
  Interventions: Drug: The combination treatment of anlotinib, penpulimab and capecitabine.

INTERVENTIONS:
Drug: The combination treatment of anlotinib, penpulimab and capecitabine. — Patients will receive the combination treatment of anlotinib, penpulimab and capecitabine every three weeks until PD or intolerance to drug toxicity. For each cycle, patients receive anlotinib 10mg, po, qd from day 1 to day 14, penpulimab 200mg, iv in day 1, and capecitabine 650mg/m2, po, bid.

SUMMARY:
First-diagnosed metastasis or recurrence/metastasis NPC Patients will be treated with anlotinib, penpulimab and capecitabine.

DETAILED DESCRIPTION:
The trial is an open-label, single-arm, phase II clinical trial. This trial plans to enroll patient that is diagnosed with locoregionally advanced nasopharyngeal carcinoma at his/her first diagnosis, and has recurrence/metastasis at least 6 months after completing radiotherapy and chemotherapy for the primary lesion, and has never accepted systemic treatment for recurrent/metastatic lesion before. The first-line treatment is the three-drug treatment plan, including anlotinib, penpulimab and capecitabine, for 4-6 cycles. Then a maintenance treatment will be run, including penpulimab and capecitabine, until PD or intolerance to toxicity.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included only when they meet all inclusion criteria.

* Between 18 to 65 years old.
* ECOG PS score 0-1 point.
* Having at least one measurable lesion confirmed by the RECIST 1.1.
* Locoregionally advanced nasopharyngeal carcinoma patients, who have never received systematic treatment for recurrent or metastatic lesion, was found with recurrence or metastasis in at least 6 months after completing chemotherapy and radiotherapy of the primary lesion. Never receive immune-checkpoint inhibitors (anti-PD-1 monoclonal antibody or anti PD-L1 monoclonal antibody, etc) treatment. In radical treatment phase of locoregional nasopharyngeal carcinoma, patients received no more than 1 type of immune-checkpoint inhibitor (limited to CTLA-4/PD-1/PD-L1 monoclonal antibody, not including bi-specific antibody or penpulimab) can be included:

  i: If the patient received immune-checkpoint inhibitors (with or without other drugs) during induction therapy, the optimal treatment effect should be PR or better than PR.

ii: If the patient received immune-checkpoint inhibitors (with or without other drugs) during radiotherapy, there should be no progression during treatment and within 6 months after treatment.

* According to the researchers' judgement, the target lesion cannot benefit from radiotherapy.
* The major organs' function is normal, and meets following criteria 7 days before intervention:

  1. Blood routine should meet (No blood transfusion or blood product within the past 14 days, and no correction was used with G-CSF or other hematopoietic stimulating factors.):

     1. Hemoglobin (HB) ≥ 90g/L;
     2. White blood cell (WBC) ≥ 4*109/L;
     3. Blood platelet (PLT): 100_109/L;
  2. Biochemistry examination should meet:

     1. Total bilirubin (TBIL) ≤ 1.5*upper limit of normal (ULN);
     2. Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5*ULN;
     3. Serum creatinine (Cr) ≤ 1.5×ULN and creatinine clearance (CCr) ≥ 60ml/min;
  3. Coagulation function: INR and APTT ≤ 1.5*ULN;
  4. Myocardial injury, heart failure three indexes examination, electrocardiogram results are normal; For patients with abnormalities in these three examinations, the researchers will assess whether to add Doppler ultrasound.
  5. Thyroid gland function: TSH ≤ ULN; If not, including those whose FT3 and FT4 levels are normal, and excluding others.
* Fertile women must already used reliable contraceptive measures or have negative gestational test (serum) result within the 7 days before inclusion. And they are willing to take suitable contraceptive measures during the clinical trial and the 8 weeks after the last administration of intervention or have sterilized. Men must take suitable contraceptive measures during the clinical trial and the 8 weeks after the last administration of intervention or have been surgically sterilized.
* Patient has signed the informed consent and has good compliance.

Exclusion Criteria:

Patients who meet any of the following criteria should be excluded:

* Disease progression within 6 months after the standard therapy of locoregional advanced nasopharyngeal carcinoma;
* Patients who cannot accept MR examination for metal implant or claustrophobia;
* Patients who need systemically using glucocorticoid (> 10mg prednisone per day) or other immunosuppressive drugs treatment in 14 days before intervention or during intervention. If the patient doesn't have active autoimmune disease, it is allowed to use invasive or topical corticosteroid and adrenocorticotropic hormone (ACTH) that is equivalent to > 10mg/day prednisone, and ACTH replacement therapy that is equivalent to ≤ 10mg/ day prednisone therapeutic dose.
* Patient who has recurrent lesion that is suitable for operation or second-course radiotherapy or, based on the judgement of the doctor in charge, can profit from the radiotherapy for the target lesion.
* Patient has active immune or autoimmune disease history, or known allograft history, or allogeneic hematopoietic stem cell transplantation history, excluding type 1 diabetes, hypothyroidism that need hormone replacement therapy and dermatologic diseases that don't need systemic treatment (e.g. leucoderma, psoriasis and alopecia.).
* Patients who had active or uncontrolled severe infection (≥ CTCAE level 3 infection) within the 4 weeks before inclusion;
* Patient who had active tuberculosis history in the past 1 year, with or without treatment. Apart from those with a proven history of regular antituberculosis therapy, patients with > 1-year active pulmonary tuberculosis history should be excluded.
* Patients with hypertension history, and their blood pressure was not well-controlled (systolic pressure ≥ 150 mmHg or diastolic pressure ≥ 90 mmHg) after 1 kind of drug treatment.
* Having significant clinical ischemia symptom or specific ischemia tendency, especially to exclude locoregional recurrent cases with high risk of ischemia;
* Urine routine examination revealed urine protein ≥ ++, and is proven that 24-h urinary protein volume ≥ 1.0g;
* Patients who had ≥ level I myocardial ischemia, myocardial infarction, arrythmia (including QTc ≥ 480ms) or ≥ level 2 congestive heart failure (New York Heart Association, NYHA) during the 6 months before inclusion.
* If the patient need Doppler ultrasound examination (the 4th of inclusion criteria 5), the abnormal result is when left ventricular ejection fraction (LVEF) < lower limit of normal (60%);
* Patient who has been diagnosed with other malignant carcinoma, excluding cured non-melanoma skin cancer, carcinoma in situ of cervix or papillary thyroid carcinoma;
* Existed meningeal metastasis or central nerve system metastasis;
* HIV positive, TP positive, liver cirrhosis, decompensated liver disease, active hepatitis (active hepatitis that were not well-controlled after treatment (Hepatitis B: HBsAg positive and HBV DNA ≥ 1*104 copies/ml; Hepatitis C: HCV RNA positive and abnormal hepatic function; the co-infection of hepatitis B and hepatitis C), and need to receive antiviral treatment;
* Patients who have participated in other anti-tumor drug-related clinical trial in the 4 weeks before inclusion;
* Patients who have received attenuated live vaccine or AK-105 treatment in the 30 days before inclusion;
* Patients who had severe hypersensitivity history to other monoclonal antibody;
* Patients who had great difficulty for oral drugs, e.g. cannot swallow, chronic diarrhea and bowel congestion, etc.
* Patients with mental drug abuse history and cannot withdrawal or mental disorder;
* There are conditions that, in the investigator's judgment, seriously endanger patient safety, may confuse the study results, or concomitant diseases or any other situations that affect the patient's completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS） | 3-year
  Progression-free survival is measured according to the RECIST 1.1.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Median value
  Objective remission rate is measured according to the RECIST 1.1.
Progression-free survival (PFS) | 3-year
  Progression-free survival is measured according to the iRECIST.
Overall survival (OS) | 3-year
  Overall survival is measured from day of diagnosis until death due to any cause or the latest known date alive.
Quality of Life (QoL) | 3-year
  Quality of Life is measured by the Quality of Life Questionnaire-Core 30 module (QLQ-C30) designed by European Organisation for Research and Treatment of Cancer (EORTC).
Quality of Life (QoL) | 3-year
  Quality of Life is measured by the FACT-H&N designed by The Center on Outcomes Research and Education.
Incidence of toxicities | 3-year
  Incidence of toxicities are measured by questionnaires covering adverse effect (AE), severe adverse effect (SAE), treatment-related adverse effect (TRAE), treatment-related severe adverse effect (TRSAE), immune-related adverse effect, immune-related treatment-related adverse effect according to NCI-CTC AE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Qu S, Li J, Hu C, Xu M, Li W, Zhou T, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Zhang W, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhang B, Yang Q, Zhang X, Zou J, Fang W, Zhang L. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1162-1174. doi: 10.1016/S1470-2045(21)00302-8. Epub 2021 Jun 23. PMID 34174189
- [Background] Cai, Q. & Su, N. & Fang, Y. & Ma, S. & Xia, Y. & Zhang, X. & Liu, P. & Yang, H.. (2020). 929P Anlotinib in patients with recurrent or metastatic nasopharyngeal carcinoma: An interim analysis of a phase II clinical trial. Annals of Oncology. 31. S668. 10.1016/j.annonc.2020.08.1044.
- [Background] Hui EP, Ma BBY, Loong HHF, Mo F, Li L, King AD, Wang K, Ahuja AT, Chan CML, Hui CWC, Wong CH, Chan ATC. Efficacy, Safety, and Pharmacokinetics of Axitinib in Nasopharyngeal Carcinoma: A Preclinical and Phase II Correlative Study. Clin Cancer Res. 2018 Mar 1;24(5):1030-1037. doi: 10.1158/1078-0432.CCR-17-1667. Epub 2018 Jan 4. PMID 29301831
- [Background] Yuan M, Zhai Y, Men Y, Zhao M, Sun X, Ma Z, Bao Y, Yang X, Sun S, Liu Y, Zhang W, Hui Z. Anlotinib Enhances the Antitumor Activity of High-Dose Irradiation Combined with Anti-PD-L1 by Potentiating the Tumor Immune Microenvironment in Murine Lung Cancer. Oxid Med Cell Longev. 2022 Feb 1;2022:5479491. doi: 10.1155/2022/5479491. eCollection 2022. PMID 35154567
- [Background] Chen YP, Liu X, Zhou Q, Yang KY, Jin F, Zhu XD, Shi M, Hu GQ, Hu WH, Sun Y, Wu HF, Wu H, Lin Q, Wang H, Tian Y, Zhang N, Wang XC, Shen LF, Liu ZZ, Huang J, Luo XL, Li L, Zang J, Mei Q, Zheng BM, Yue D, Xu J, Wu SG, Shi YX, Mao YP, Chen L, Li WF, Zhou GQ, Sun R, Guo R, Zhang Y, Xu C, Lv JW, Guo Y, Feng HX, Tang LL, Xie FY, Sun Y, Ma J. Metronomic capecitabine as adjuvant therapy in locoregionally advanced nasopharyngeal carcinoma: a multicentre, open-label, parallel-group, randomised, controlled, phase 3 trial. Lancet. 2021 Jul 24;398(10297):303-313. doi: 10.1016/S0140-6736(21)01123-5. Epub 2021 Jun 7. PMID 34111416
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Background] Wang X, Teng F, Kong L, Yu J. PD-L1 expression in human cancers and its association with clinical outcomes. Onco Targets Ther. 2016 Aug 12;9:5023-39. doi: 10.2147/OTT.S105862. eCollection 2016. PMID 27574444
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405